CLINICAL TRIAL: NCT04959500
Title: Addition of Anlotinib Hydrochloride to the Stupp Regimen Versus the Stupp Regimen Alone for Newly Diagnosed Glioblastoma: A Randomized Double-blind Multicenter Prospective Phase II Study
Brief Title: Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhongping Chen, clinical professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-Ⅱ-01
Record Dates: First submitted 2021-06-23; First posted 2021-07-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental: Radiation therapy, Temozolomide and anlotinib Patients will receive standard radiation therapy plus temozolomide (Stupp regimen). Anlotinib hydrochloride will be given with a daily dose of 10 mg for 14 days of a 21-day cycle up to 2 cycles, initiated on the first day of radiation therapy and followed by adjuvant treatment with the same dosing schedule until patients have disease progression or intolerable toxicities.
  Interventions: Drug: Anlotinib Hydrochloride; Radiation: Radiation Therapy; Drug: Temozolomide
- control group (Placebo Comparator): Experimental: Radiation therapy, Temozolomide and Placebo Patients will receive standard radiation therapy plus temozolomide (Stupp regimen). Placebo will be given with a daily dose of 0 mg for 14 days of a 21-day cycle up to 2 cycles, initiated on the first day of radiation therapy and followed by adjuvant treatment with the same dosing schedule until patients have disease progression or intolerable toxicities.
  Interventions: Drug: Placebo; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Drug: Anlotinib Hydrochloride Anlotinib hydrochloride will be given with a daily dose of 12 mg for 14 days of a 21-day cycle up to 2 cycles, initiated on the first day of radiation therapy and followed by adjuvant treatment with the same dosing schedule until patients have disease progression or intolerable toxicities.
  Arms: Experimental group
Drug: Placebo — Drug: Placebo Placebo will be given with a daily dose of 12 mg for 14 days of a 21-day cycle up to 2 cycles, initiated on the first day of radiation therapy and followed by adjuvant treatment with the same dosing schedule until patients have disease progression or intolerable toxicities.
  Arms: control group
Radiation: Radiation Therapy — Radiation: Radiation therapy Radiation therapy will be delivered in daily fractions of 1.8-2.0 Gy given 5 days a week for a total of 54-60 Gy.
Drug: Temozolomide — Drug: Temozolomide Temozolomide will be administered at a daily dose of 75 mg/m2 until the completion of radiation therapy. Four weeks after the completion of radiation therapy, patients will be given with adjuvant chemotherapy with temozolomide at a dose of 200 mg/m2 for 5 days of a 28-day cycle for a total of 6 cycles.

SUMMARY:
Addition of Anlotinib Hydrochloride to the Stupp Regimen Versus the Stupp Regimen Alone for Newly Diagnosed Glioblastoma.Take PFS as the main evaluation index, the purpose is to evaluate its effectiveness

ELIGIBILITY:
Inclusion Criteria:

* Understood and Signed an informed consent form., with good compliance
* Age: 18-75 years old；.Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2；Life expectancy of at least 3 months.
* Glioblastoma confirmed by histology ;
* Random time is 4-6 weeks from the last operation , and the investigator judges that the surgical wound has healed well;
* Within 5 days before administration, the dosage of corticosteroids was stable or gradually decreased;
* Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study ；Not Pregnant or breastfeeding women,Pregnancy before pregnancy screening, the women who blood / urine results were positivetherapy.

Exclusion Criteria:

* Have previously received systemic radiotherapy and chemotherapy for GBM;
* IDH1/2 mutations are present
* Contraindicated for MRI examination
* The tumor only occurs in the brain stem
* Radiologically obvious diffuse meningeal dissemination
* Imaging shows that the tumor has invaded the periphery of important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels and cause fatal hemorrhage, cerebrovascular malformations or other bleeding tendency during the subsequent study period;
* Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident , deep vein thrombosis and pulmonary embolism；
* Other malignant tumors have occurred or are currently present at the same time within 3 years.
* There are many factors that affect oral medications ;
* Received anti-tumor Chinese patent medicine which were approved by NMPA Within 2 weeks before the start of the study.
* A clear history of neurological or psychiatric diseases, moderate or higher epilepsy , moderate or higher aphasia or dementia
* Participated in other anti-tumor drug clinical trials within 4 weeks before grouping;
* Other conditions which are not fit for this study assessed by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by IRC | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events: objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
The progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events: objective disease progression or death due to any cause.
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  OS was defined as the time from the date of study enrollment to the date of death due to any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongping Chen, Doctor, Principal Investigator — Sun Yat-sen University
Locations (22):
- China (22):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Beijing TianTan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The Sixth Madical Center of PLA General Hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army (PLAGH), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The Fifth Affiliated Hospital Sun Yat-sen University, Zhuhai, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The affiliated hospital of xuzhou medical university, Xuzhou, Jiangsu
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Gansu Provincial Hospital, Gansu, Lanzhou Province
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University shabghai cancer center, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of PLA Air Force Medical University, Xian, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang